CLINICAL TRIAL: NCT02030639
Title: Phase I Study of the Metabolism and Excretion of [14C]-Rigosertib After Single-dose Administration as 24-hour Continuous Intravenous Infusion to Healthy Volunteers
Brief Title: Metabolism and Excretion of [14C]-Rigosertib After Infusion to Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Onconova 04-23; 8287875 (Other: Covance Clinical Research Unit, Inc.)
Record Dates: First submitted 2014-01-07; First posted 2014-01-08 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Healthy
MeSH Terms: interventions — ON 01910

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [14C]-rigosertib (Experimental): A single dose of 450 mg of rigosertib containing 250 microcuries of carbon 14-labeled rigosertib ([14C]-rigosertib) administered as a continuous intravenous (CIV) infusion over 24 hours to healthy volunteers.
  Interventions: Drug: rigosertib

INTERVENTIONS:
Drug: rigosertib — A single dose of 450 mg of rigosertib containing 250 microcuries of carbon 14-labeled rigosertib ([14C]-rigosertib) administered as a continuous intravenous (CIV) infusion over 24 hours to healthy volunteers.
  Other Names: rigosertib sodium; ON 01910.Na

SUMMARY:
The purpose of this study is to gain an understanding of how the experimental anti-cancer drug, rigosertib, is metabolized in the body and excreted in the urine and feces after it is given as an intravenous infusion. In addition, the study will be carefully monitored to see if any side effects occur.

A radioactive drug is used in this study because it is easier and more accurate to measure radioactivity than to use more complicated and less sensitive chemical tests for the drug.

DETAILED DESCRIPTION:
This study will be an open-label, non-randomized, metabolism and excretion study of [14C]-rigosertib administered as a single dose of approximately 450 mg containing 250 μCi [14C]-labeled rigosertib as a 24-hour continuous intravenous (CIV) infusion in healthy volunteers. Up to 8 subjects will be enrolled to ensure at least 6 subjects have evaluable data.

Eligible subjects will be confined at the clinical site from the time of Check-in (approximately 24 hours prior to dosing) until Discharge (between Days 6 and 10). One single dose of [14C]-rigosertib will be administered as a 24-hour continuous intravenous infusion on Day 1. Subjects will be discharged as early as 120 hours after the start of the infusion, after ≥ 90% of the administered radioactive dose has been recovered in urine and feces or when the combined total radioactivity recovered in urine and feces is ≤ 1% of the administered radioactive dose for 2 consecutive 24-hr samples. The maximum stay will be until Day 10 (216 hours after the start of the infusion).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 kg/m2 and 29.9 kg/m2, inclusive;
* In good health, as defined by the absence of clinically significant findings from medical history, 12-lead electrocardiogram (ECG), and vital signs;
* Clinical laboratory evaluations that are within the normal range, unless deemed not clinically significant by the Investigator. Platelet (PLT) count, white blood cell (WBC) count, and absolute neutrophil count (ANC) should all be above the lower limit of normal (LLN);
* Negative test for selected drugs of abuse at Screening (does not include alcohol) and at Check-in (does include alcohol);
* Negative hepatitis panel (including hepatitis B surface antigen [HBsAg] and hepatitis C virus antibody [anti-HCV]) and negative human immunodeficiency virus (HIV) antibody screens;
* Males will either be vasectomized or sterile;
* Female subjects must have undergone confirmed tubal ligation or hysterectomy or be post-menopausal;
* Able to comprehend and willing to sign an informed consent form (ICF);
* History of a minimum of 1 bowel movement per day.

Exclusion Criteria:

* Participation in any other investigational study drug trial in which receipt of an investigational agent, biologic agent, small targeted molecule, or immunotherapy occurred within 5 half-lives or 4 weeks of enrollment, whichever is longer;
* Major surgery within 3 weeks of enrollment or major surgery without full recovery;
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs except that appendectomy and hernia repair will be allowed;
* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder;
* History of Gilbert's Syndrome;
* History or presence of an abnormal ECG, which, in the Investigator's opinion, is clinically significant;
* Uncontrolled hypertension, defined as systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg, unless deemed acceptable by the Investigator;
* History of seizures, except febrile seizures as a child;
* Psychiatric illness/social situations that would limit the subject's ability to tolerate and/or comply with study requirements, or inability to comply with study and/or follow-up procedures;
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator;
* History of alcoholism or drug addiction within 1 year prior to Check-in;
* Participation in more than 1 other radiolabeled investigational study drug trial within 12 months prior to Check-in. The previous radiolabeled study drug must have been received more than 6 months prior to Check-in for this study and the total exposure from this study and the previous study will be within the recommended levels considered safe;
* Exposure to significant radiation within 12 months prior to Check-in;
* Use of any prescription medications/products within 14 days prior to Check-in, unless deemed acceptable by the Investigator;
* Use of any over-the-counter, non-prescription preparations within 7 days prior to Check-in, unless deemed acceptable by the Investigator;
* Poor peripheral venous access;
* Donation of blood from 30 days prior to Screening through discharge, inclusive, or of plasma from 2 weeks prior to Screening through discharge, inclusive;
* Receipt of blood products within 2 months prior to Check-in;
* Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The mean percent of the radioactivity of the administered doses recovered in the urine, feces, and overall (urine + feces) | Up to 216 hours
  Urine sample collection for radio analysis will be over the intervals of 24-30 hours (hr), 30-36 hr, 36-42 hr, 42-48 hr, 48-72 hr, 72-96 hr, 96-120 hr, and if necessary based on discharge criteria, at 120-144 hr, 144-168 hr, 168-192 hr, and 192-216 hr after the infusion start. Fecal sample collection for radio analysis will be over the intervals of 24-30 hr, 30-36 hr, 36-42 hr, 42-48 hr, 48-72 hr, 72-96 hr, 96-120 hr, and if necessary based on discharge criteria, at 120-144 hr, 144-168 hr, 168-192 hr, and 192-216 hr after the infusion start.
Concentration of rigosertib in plasma | Up to 216 hours
  Concentration of rigosertib in plasma will be measured by a validated high performance liquid chromatography (HPLC) method. Plasma samples will be collected at 24 hours (hr) (immediately before the end of the infusion), 24.25 hr, 24.5 hr, 25 hr, 26 hr, 28 hr, 30 hr, 36 hr, 48 hr, 72 hr, and 96 hr after the infusion start, and, if the subject has not been discharged by then, at 144 hr, 192 hr, and 216 hr after the infusion start. Concentration values will be used to derive the following pharmacokinetic parameters: Cmax; tmax; AUC0-t; AUC0-∞; λZ; t1/2; CL; Vz; Vss.
Concentration of radioactivity in whole blood | Up to 216 hours
  Blood samples for radio analysis will be collected at 24 hours (hr) (immediately before the end of the infusion), 24.25 hr, 24.5 hr, 25 hr, 26 hr, 28 hr, 30 hr, 36 hr, 48 hr, 72 hr, and 96 hr after the infusion start, and, if the subject has not been discharged by then, at 144 hr, 192 hr, and 216 hr after the infusion start.
Concentration of radioactivity in plasma | Up to 216 hour
  Plasma samples for radio analysis will be collected at 24 hours (hr) (immediately before the end of the infusion), 24.25 hr, 24.5 hr, 25 hr, 26 hr, 28 hr, 30 hr, 36 hr, 48 hr, 72 hr, and 96 hr after the infusion start, and, if the subject has not been discharged by then, at 144 hr, 192 hr, and 216 hr after the infusion start.

SECONDARY OUTCOMES:
Metabolite profiling | Up to 216 hours
  Extracts from samples of plasma, urine and feces will be subjected to high performance liquid chromatography (HPLC) with radiochemical detection for the quantitative analysis of rigosertib and its metabolites.
Metabolite identification | Up to 216 hours
  Metabolite identification will be carried out by mass spectrometry. Synthetic standards of known metabolites will be used to confirm identifications.
Concentration of radioactivity in urine | Up to 216 hours
  Urine sample collection for radio analysis will be over the intervals of 24-30 hr, 30-36 hr, 36-42 hr, 42-48 hr, 48-72 hr, 72-96 hr, 96-120 hr, and if necessary based on discharge criteria, at 120-144 hr, 144-168 hr, 168-192 hr, and 192-216 hr after the infusion start.
Concentration of radioactivity in feces | Up to 216 hours
  Fecal sample collection for radio analysis will be over the intervals of 24-30 hr, 30-36 hr, 36-42 hr, 42-48 hr, 48-72 hr, 72-96 hr, 96-120 hr, and if necessary based on discharge criteria, at 120-144 hr, 144-168 hr, 168-192 hr, and 192-216 hr after the infusion start.
Number of subjects who experience an adverse event | Up to 31 days
  An adverse event is defined according to ICH E2A guidance.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Wilhelm, MD, PhD, Study Chair — Traws Pharma, Inc.
Locations (1):
- Covance Clinical Research Unit, Inc., Madison, Wisconsin, United States

REFERENCES:
- [Result] Garcia-Manero G, Fenaux P. Comprehensive Analysis of Safety: Rigosertib in 557 Patients with Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML). Blood Dec 2016, 128 (22) 2011; ASH 2016.